CLINICAL TRIAL: NCT06873984
Title: Compression Stockings for Preventing Lower Limb Lymphedema in Women Treated for Gynecological Malignancies
Brief Title: Compression Stockings for Lymphedema Prevention in Gynecologic Cancer Patients
Acronym: csplwgm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joanna Kurpiewska-Pieniążek (Other)
Responsible Party: Sponsor-Investigator, Joanna Kurpiewska-Pieniążek, Principal Investigator, PhD, Andrzej Frycz Modrzewski Krakow University
Organization: Andrzej Frycz Modrzewski Krakow University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Csplwgm-AFMKU
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Lymphedema
Keywords: Lower limb lympodema, compression therapy, quality of life
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compression Group (CG) (Experimental): Experimental: Compression Group (CG) Women in the CG group were provided with individually fitted round-knit compression stockings with a pressure of 23-32 mmHg (class 2, RAL-GZG standard classification). They received detailed instructions on usage, recommending approximately 9 hours of wear per day. The compression garments were selected based on circumference measurements taken in the morning and were sourced from the same manufacturer (Medi GmbH & Co., Bayreuth, Germany).
  In addition, physical activity (PA) was encouraged, specifically walking for 20 minutes daily, with compression stockings worn during the activity. All participants received comprehensive education on skin care, self-manual lymph drainage (simple lymph drainage, SLD), and lymphedema prevention. Proper skin hygiene was maintained through daily washing with hypoallergenic soap, thorough drying (especially between the toes and fingers), and regular skin moisturizing. A simplified version of manual lymph drainage wa
  Interventions: Other: compression products
- No Compression Group (NCG) (No Intervention): Women in the NCG group did not receive compression therapy. However, they were encouraged to :
  Physical activity (PA) was recommended, specifically walking for 20 minutes every day.
  All women received comprehensive education on skin care, self-manual lymph drainage (simple lymph drainage, SLD), and lymphedema prevention. Proper skin hygiene was maintained through daily washing with hypoallergenic soap, thorough drying (especially between the fingers), and regular skin moisturizing.
  A simplified version of manual lymph drainage aimed at improving lymphatic flow was recommended for 20 minutes per day. The technique included the unaffected areas of the body (neck, chest, and abdomen).

INTERVENTIONS:
Other: compression products — Compression Group (CG):
  Participants received individually fitted, round-knit compression stockings with a pressure of 23-32 mmHg (Class 2, RAL-GZG standard).
  Compression garments were selected based on circumference measurements taken in the morning to ensure proper fit.
  Participants were instructed to wear the stockings for approximately 9 hours per day.
  The compression garments were provided by the same manufacturer (Medi GmbH & Co., Bayreuth, Germany).
  Additionally, participants were advised to engage in daily physical activity (walking for at least 20 minutes per day) while wearing compression.
  Comprehensive education was provided on skin care, self-manual lymph drainage (simple lymph drainage, SLD), and lymphedema prevention.
  Arms: Compression Group (CG)

SUMMARY:
The goal of this clinical trial was to evaluate whether compression stockings (23-32 mmHg) reduce the incidence of postoperative lymphedema and accompanying symptoms, as well as to assess the comfort of using compression in women undergoing treatment for gynecological malignancies up to one year after surgery.

The main objectives were to determine:

Whether compression stockings applied immediately after radical surgery, in combination with physical activity, reduce the risk of developing lymphedema.

Whether the use of compression stockings affects the quality of life. Whether compression stockings influence specific physical complaints related to the lower limbs.

Patients were assessed preoperatively and at 3, 6, and 12 months postoperatively. Limb circumferences were measured at predefined anatomical points to calculate limb volume changes over time. Additionally, subjective symptoms, quality of life, and adherence to compression therapy were evaluated.

Researchers compared a group using compression stockings with a control group without compression to analyze potential benefits and complications.

DETAILED DESCRIPTION:
Background and Rationale Lymphedema is a frequent and debilitating complication following radical surgery for gynecological malignancies. It affects patients' quality of life, contributing to discomfort, impaired mobility, and an increased risk of infections. Despite the widespread use of compression therapy in managing lymphedema, there is limited evidence on its preventive role when applied immediately after surgery.

This study investigates the effectiveness of compression stockings (23-32 mmHg) in reducing the incidence of postoperative lower limb lymphedema and associated symptoms in women undergoing treatment for gynecological cancers. Additionally, it evaluates the impact of compression on patients' quality of life and physical complaints up to one year postoperatively.

A total of 75 eligible women consented to participate and were preoperatively randomized (simple randomization using a random number generator) into two groups:

Compression Group (CG): Patients received individually fitted round-knit compression stockings (23-32 mmHg, RAL-GZG standard) and were instructed to wear them for approximately 9 hours per day.

No Compression Group (NCG): Patients did not receive compression therapy.

Descriptive statistics were used to summarize the collected data, including mean (x̄), standard deviation (SD), median (Me), and percentage distributions.

For sociodemographic and clinical data, comparisons between groups were performed using the chi-square test for categorical variables and the independent t-test for continuous variables.

The effects of physiotherapeutic interventions were analyzed to determine statistically significant differences between groups. To assess the normality of data distribution, the Shapiro-Wilk test was applied.

For quantitative variables related to limb volume and WAC (Water-Assisted Circumference), comparisons between two groups were conducted using the Mann-Whitney U test. Comparisons of quantitative variables across three or more groups were performed using the Kruskal-Wallis test, followed by Dunn's post-hoc test when significant differences were detected.

Correlations between quantitative variables (e.g., limb volume and WAC) were assessed using Spearman's correlation coefficient.

For repeated measurements of quantitative variables (e.g., limb volume and WAC at multiple time points), comparisons were conducted using the Friedman test, and when significant differences were found, Wilcoxon signed-rank tests with Bonferroni correction were used for post-hoc analysis.

Qualitative variables were analyzed by calculating the number and percentage of occurrences for each category. Comparisons of categorical variables between groups were performed using the chi-square test (with Yates' correction for 2x2 tables) or Fisher's exact test for small expected frequencies.

For comparisons of continuous variables across two time points, the Wilcoxon signed-rank test for paired samples was used.

A significance level of p < 0.05 was adopted, and all p-values below this threshold were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Women who underwent radical surgery for vulvar cancer. Women who underwent radical surgery for cervical, uterine, or ovarian cancer, with systemic pelvic lymph node dissection.

Overweight or obese patients (BMI > 25.0 kg/m²) treated for uterine or ovarian cancer, regardless of whether systemic pelvic lymph node dissection was performed.

Women over 18 years of age.

Exclusion Criteria:

Women with a history of lymphedema, venous edema, an ECOG score > 2, congestive heart failure, renal failure, hypothyroidism, leg ulcers, or severe lower limb ischemia (Fontaine class ≥ 2), as well as those with metastases, relapse, or other malignancies treated within five years prior to study entry, were excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Lower Limb Volume (%) | Measurements were taken preoperatively and at 3, 6, and 12 months postoperatively
  Lower limb volume change (%) was calculated based on circumferential measurements taken every 4 cm along the limb, using the truncated cone formula. . The percentage change was calculated relative to preoperative limb volume.
  Unit of Measure: Percentage (%)

SECONDARY OUTCOMES:
Presence of Lymphedema | were noted before and after 3, 6 and 12 months after surgery
  Description: Lymphedema was diagnosed if limb volume increased by ≥10% compared to the contralateral limb or if skin stiffness appeared with a ≥8% volume difference.
  Unit of Measure: Number of participants with lymphedema
Relative Edema Size (%) | were taken before and after 3, 6 and 12 months after surgery i
  If edema occurred, its relative size (%) was calculated as the volume difference between the affected and healthy limb, expressed as a percentage of the healthy limb's volume.
  Unit of Measure: Percentage (%)
Weight-Adjusted Volume Change (WAC) (%) | were taken before and after 3, 6 and 12 months after surgery
  To account for body weight fluctuations, limb volume was normalized using the WAC formula:
  WAC = (A2 * W1) / (W2 * A1) - 1 where A1 and A2 were pre- and postoperative limb volumes, and W1 and W2 were pre- and postoperative body weights.
  Unit of Measure: Percentage (%)

OTHER OUTCOMES:
Physical Symptoms Related to Lower Limb Lymphedema | Symptoms were recorded before surgery and at 3, 6, and 12 months postoperatively.
  The frequency of six physical symptoms associated with lower limb lymphedema (pain, limb heaviness, skin tightness, numbness, genital swelling, and lymph leakage) was assessed using a custom Likert-type scale (0 = never, 1 = sometimes, 2 = often, 3 = very often, 4 = all the time). Participants rated these symptoms preoperatively and at 3, 6, and 12 months post-treatment.
  Unit of Measure: Likert scale score (0-4)
The assessment of compression compliance | 12 months postoperatively
  was based on the International Compression Questionnaire (ICC) taking into account the functional condition of women before starting to use compression and the evaluation of the tested compression stockings after 12 months in CG group. The severity of physical conditions reported before beginning to use compression was presented on a numeric rating scale (NRS) from 0 to 10, where 0 denoted no symptoms and 10 stood for a very high severity of a given symptom.
  Compression comfort (easy donning; easy doffing; feeling immediately after donning; feeling during daytime; putting on clothes on compression; the appearance of the garment (NRS: 0 = not able at all, 10 = completely able, sum of points) and complications of compression related to skin irritation, tender, spots. skin damage, itching, warmth, throbbing, cramps, cutting in, slippage, local swelling, bulky feeling, and too-tight feeling (NRS: 0 = not present at all, 10 = very obviously present
Quality of Life (EORTC QLQ-C30 Score) | Assessments were conducted at 12 months postoperatively
  Quality of life was assessed using the standardized EORTC QLQ-C30 (version 3.0) questionnaire for cancer patients. It included five functional scales (physical, role, emotional, cognitive, and social functioning), three symptom scales (fatigue, nausea/vomiting, pain), six single-item symptom questions (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties), and two global health status questions. Scores were analyzed according to EORTC scoring guidelines.
  Unit of Measure: EORTC QLQ-C30 score (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kurpiewska-Pieniążek, PhD, Principal Investigator — Andrzej Frycz Modrzewski Krakow University, Krakow, Poland
Locations (2):
- Poland (2):
  - Clinical Department of Gynecology and Gynecologic Oncology, University Hospital in Krakow"., Krakow, Lesser Poland Voivodeship
  - Department of Gynecology and Obstetrics, including Gynecologic Oncology, Krakow, Lesser Poland Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ochalek K, Gradalski T, Partsch H. Preventing Early Postoperative Arm Swelling and Lymphedema Manifestation by Compression Sleeves After Axillary Lymph Node Interventions in Breast Cancer Patients: A Randomized Controlled Trial. J Pain Symptom Manage. 2017 Sep;54(3):346-354. doi: 10.1016/j.jpainsymman.2017.04.014. Epub 2017 Aug 8. PMID 28797867
- [Background] Stuiver MM, de Rooij JD, Lucas C, Nieweg OE, Horenblas S, van Geel AN, van Beurden M, Aaronson NK. No evidence of benefit from class-II compression stockings in the prevention of lower-limb lymphedema after inguinal lymph node dissection: results of a randomized controlled trial. Lymphology. 2013 Sep;46(3):120-31. PMID 24645535
- [Background] Sawan S, Mugnai R, Lopes Ade B, Hughes A, Edmondson RJ. Lower-limb lymphedema and vulval cancer: feasibility of prophylactic compression garments and validation of leg volume measurement. Int J Gynecol Cancer. 2009 Dec;19(9):1649-54. doi: 10.1111/IGC.0b013e3181a8446a. PMID 19955953
- [Background] Hsu YY, Liu CY, Ho CL, Hsu KF. Determinants of quality of life related to lower limb lymphedema in women with gynecological cancer surgery. Asia Pac J Oncol Nurs. 2022 Oct 3;10(1):100153. doi: 10.1016/j.apjon.2022.100153. eCollection 2023 Jan. PMID 36406465
- [Background] Bowman C, Piedalue KA, Baydoun M, Carlson LE. The Quality of Life and Psychosocial Implications of Cancer-Related Lower-Extremity Lymphedema: A Systematic Review of the Literature. J Clin Med. 2020 Oct 2;9(10):3200. doi: 10.3390/jcm9103200. PMID 33023211
- [Background] Russo S, Walker JL, Carlson JW, Carter J, Ward LC, Covens A, Tanner EJ 3rd, Armer JM, Ridner S, Hayes S, Taghian AG, Brunelle C, Lopez-Acevedo M, Davidson BA, Schaverien MV, Ghamande SA, Bernas M, Cheville AL, Yost KJ, Schmitz K, Coyle B, Zucker J, Enserro D, Pugh S, Paskett ED, Ford L, McCaskill-Stevens W. Standardization of lower extremity quantitative lymphedema measurements and associated patient-reported outcomes in gynecologic cancers. Gynecol Oncol. 2021 Feb;160(2):625-632. doi: 10.1016/j.ygyno.2020.10.026. Epub 2020 Nov 4. PMID 33158510
- [Background] Huang J, Yu N, Wang X, Long X. Incidence of lower limb lymphedema after vulvar cancer: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Nov;96(46):e8722. doi: 10.1097/MD.0000000000008722. PMID 29145314
- [Background] Yoshihara M, Shimono R, Tsuru S, Kitamura K, Sakuda H, Oguchi H, Hirota A. Risk factors for late-onset lower limb lymphedema after gynecological cancer treatment: A multi-institutional retrospective study. Eur J Surg Oncol. 2020 Jul;46(7):1334-1338. doi: 10.1016/j.ejso.2020.01.033. Epub 2020 Jan 31. PMID 32146054
- [Background] Wu X, Liu Y, Zhu D, Wang F, Ji J, Yan H. Early prevention of complex decongestive therapy and rehabilitation exercise for prevention of lower extremity lymphedema after operation of gynecologic cancer. Asian J Surg. 2021 Jan;44(1):111-115. doi: 10.1016/j.asjsur.2020.03.022. Epub 2020 May 10. PMID 32402630
- [Background] Hayes SC, Janda M, Ward LC, Reul-Hirche H, Steele ML, Carter J, Quinn M, Cornish B, Obermair A. Lymphedema following gynecological cancer: Results from a prospective, longitudinal cohort study on prevalence, incidence and risk factors. Gynecol Oncol. 2017 Sep;146(3):623-629. doi: 10.1016/j.ygyno.2017.06.004. Epub 2017 Jun 16. PMID 28624154
- See also: This page provides detailed information about the EORTC QLQ-C30 questionnaire, a standardized tool used to assess the quality of life in cancer patients. — https://www.eortc.org/
- See also: Postoperative Effectiveness of Comprehensive Nursing Intervention for Lymphedema in Gynecological Cancer: A Controlled Study — https://pubmed.ncbi.nlm.nih.gov/37295012/
- See also: International Society of Lymphology — https://www.lk-lymphoedema.com/2010/03/international-society-of-lymphology/